CLINICAL TRIAL: NCT06971965
Title: Necessity of TSH Suppression Therapy in Active Surveillance for Thyroid Cancer Patients.
Acronym: MAeSTro-TSH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0173
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer; Papillary Thyroid Carcinoma
Keywords: Active Surveillance
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low TSH group (Experimental): 0.3 ≤ target TSH <2.0mIU/L
  Interventions: Drug: Levothyroxin
- high TSH group (Experimental): 2.0 ≤ target TSH <8.0mIU/L
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Levothyroxin — During the five-year study intervention period, thyroid hormone (oral administration) supplementary doses are determined according to a dose-adjustment protocol established for the group's target TSH range.

SUMMARY:
This study is a multicenter randomized controlled trial conducted in Korea. A parallel, two-group randomized design will be with thyroid stimulating hormone suppression therapy group(low TSH group; intervention) is different from the wIthout thyroid stimulating hormone (TSH) suppression therapy group(high TSH group; control).

DETAILED DESCRIPTION:
Patients diagnosed with papillary thyroid cancer who wanted Active surveillance and meet the inclusion / exclusion criteria will be randomized 1: 1 into two groups: the high TSH and low TSH group. During the study period, thyroid hormone supplementary doses will be determined according to the dose-adjustment protocol established for each target TSH range.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule of 1.0 cm or less confirmed as Bethesda category V (suspicious for PTC) or VI (PTC) based on cytopathological examination, or Bethesda category III (atypia of undetermined significance) with a confirmed BRAF V600E mutation.
* Patients with no evidence of distant metastasis, cervical lymph node metastasis, recurrent laryngeal nerve invasion, or tracheal invasion. Additionally, no evidence of extrathyroidal extension (ETE) should be present, and the tumor must not belong to high-risk subtypes of PTC (e.g., diffuse sclerosing, columnar cell, or solid subtype).
* Non-pregnant women of childbearing potential (confirmed by medical history taking)

Exclusion Criteria:

* Hyperthyroidism
* If the investigator determines that you are not suitable for clinical research participation considering the following comorbidities:

  * Myocardial infarction or cerebrovascular accident within the last three months.
  * Diseases with limited life expectancy or potentially impairing the patient's ability to comply with at least five years of treatment or follow-up.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Disease progression | at 3,5years after enrollment
  The rate of disease progression will be assessed as the proportion (%) of patients with biopsy-confirmed recurrence, based on suspicious findings identified through thyroid (neck) ultrasound performed at 6- to 12-month intervals.

SECONDARY OUTCOMES:
Disease free survival | at 3,5years after enrollment
  As the time interval from enrollment to either disease progression or all-cause mortality, whichever occurs first.
Disease specific survival | at 3,5years after enrollment
  As the time from the date of enrollment to disease-specific mortality.
Overall Survival | at 3,5years after enrollment
  As the time from the date of enrollment to death.
Target-TSH-level achievement rate | at 3,5years after enrollment
  Comparison of between the low-TSH and high-TSH groups at each follow-up visit regarding the presence or absence of thyroid hormone use and its dosage, considering body weight and medication adherence, in order to achieve the target TSH concentration.
Incidence of complications | at 3,5years after enrollment
  Comparison of the incidence of complications at each follow-up visit between the low-TSH and high-TSH groups.
Safety evaluation | at 3,5years after enrollment
  Incidence and grade of adverse events.
Risk Factors for Thyroid Cancer Recurrence | at 3,5years after enrollment
  The study will assess the relationship between thyroid hormone levels (TSH, free T4, total T3 or free T3) and potential risk factors for recurrence, including:
  * Demographic factors: sex, age, smoking status, BMI
  * Pathologic features: tumor stage, size, extrathyroidal extension
  * Genetic mutations: BRAF, TERT promoter mutations
  The analysis will identify factors, adjusted for thyroid hormone levels, significantly associated with recurrence risk. Statistical methods such as Generalized Estimating Equations (GEE), Interval Censored Survival Analysis, and Cox-proportional hazards regression will be used for evaluation.
Predictors of Treatment-Related Complications Based on Thyroid Hormone Levels | at 3,5years after enrollment
  The study will assess the relationship between thyroid hormone levels (TSH, free T4, total T3 or free T3) and risk factors for treatment-related complications (e.g., tachycardia, reduced bone mineral density). Risk factors include:
  * Demographic factors: sex, age, smoking, BMI, weight, blood pressure, concurrent medications, menopausal status, diabetes, asthma/COPD, rheumatic diseases
  * Cholesterol levels: Total cholesterol, LDL, HDL
  * ECG and Bone Mineral Density (BMD)
  The analysis will evaluate the association between these factors and treatment-related complications, adjusting for thyroid hormone levels. Incidence rates of complications at follow-up will be compared using Chi-square, Fisher's exact test, or Generalized Estimating Equations (GEE).
Predictors of TSH levels and proper thyroid hormone dosage | at 3,5years after enrollment
  This study will identify factors that predict changes in thyroid hormone levels (TSH, free T4, total T3, or free T3) and predict the required thyroid medication dosing. The factors under include:
  * Demographic Factors: Sex, age, comorbidities, smoking status, body mass index (BMI), weight, and current medications
  * Thyroid Function: Pre-existing thyroid disorders, and the presence of thyroiditis
  The analysis will evaluate the association between these factors and changes in thyroid hormone levels, as well as predict the necessary adjustments in thyroid hormone dosing, using multiple regression analysis.
Test interval for efficient diagnosis of recurrence | at 3,5years after enrollment
  To analyze the duration until recurrence and the interval between examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kyung Lee, Principal Investigator — National Cancer Center; Young Joo Park, Principal Investigator — Seoul National University Hospital; Minjoo Kim, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No